CLINICAL TRIAL: NCT06364787
Title: The Safety and Efficacy Assessment of Allogeneic γδ T Cells Combined With Targeted Therapy and Immunotherapy in Hepatocellular Carcinoma Patients
Brief Title: Allogeneic Gamma-delta T Cells Combined With Targeted Therapy and Immunotherapy in a Phase 1 Clinical Trial for First-line Treatment of Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); Beijing GD Initiative Cell Therapy Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDT-001-07-01
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- γδ T cells+ PD-1 monoclonal antibody+ targeted drugs (Experimental): Patients will receive 4 cycles of ex-vivo expanded allogeneic γδ T cells treatments, at three-weeks' intervals. Ex-vivo expanded γδ T cells are transfused to patients in a typical 3+3 dose-escalation design (Dose escalation, 1×10^8/kg, 2×10^8/kg,4×10^8/kg).
  Interventions: Biological: γδ T cells; Drug: Targeted drugs; Drug: PD-1 monoclonal antibody
- PD-1 monoclonal antibody+ targeted drugs (Active Comparator): PD-1 monoclonal antibody+ targeted drugs
  Interventions: Drug: Targeted drugs; Drug: PD-1 monoclonal antibody

INTERVENTIONS:
Biological: γδ T cells — Cells will be extracted from a healthy donor by apheresis, followed by ex-vivo expansion and activation. The ex-vivo expanded γδ T cells from donors will be adoptively transfused.
  Arms: γδ T cells+ PD-1 monoclonal antibody+ targeted drugs
Drug: Targeted drugs — Multi-target kinase inhibitors can act on VEGFR-1,VEGFR-2,VEGFR-3,FGFR1,PDGFR,cKit,Ret and other targets.
Drug: PD-1 monoclonal antibody — Humanized programmed death receptor (PD-1) monoclonal antibody that binds to PD- and prevents binding of PD-1 with programed death ligands 1 (PD-L1) and PD-L2. It can function to activate cytotoxic T lymphocytes and inhibit tumor growth.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of allogeneic γδ T cells combined with targeted therapy and PD-1 monoclonal antibody in first-line treatment of patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
This is a double-arm, single-center, randomized, open label phase I clinical trial to evaluate the efficacy and safety of the combination of ex-vivo expanded allogeneic γδ T cells plus targeted therapy and PD-1 monoclonal antibody in patients with BCLC stage B or C hepatocellular carcinoma (HCC). A typical 3+3 dose-escalation design will be used to determine the optimal dose level of γδ T cells based on the incidence of dose-limiting toxicity (DLT). The initial infusion dose level will start from 1×10^8/kg to 4×10^8/kg in every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should sign informed consent form voluntarily before the trail and comply with the requirements of this study.
2. Age 18 years up to the age of 75 (≤75), gender unlimited.
3. Hepatocellular Carcinoma diagnosed according to the 2018 edition of the EASL guidelines.
4. BCLC stage B or C.
5. Liver function: Child-Pugh class A/B (5-9).
6. Eastern Cooperative Oncology Group (ECOG) Performance score≤1.
7. No previous antitumor therapy.
8. Life expectancy ≥ 6 months.
9. Patients combined with HBV infection require antiviral treatment with nucleoside analogues; patients combined with HCV infection require direct-acting antiviral agent (DAA) treatment.
10. Adequate organ and marrow function (within 4 weeks prior to study treatment initiation).
11. Male and female patients of reproductive potential must agree to use birth control during the study and for at least 30 days post study.
12. Capable of understanding and complying with the study protocol requirements ( including follow-up visit and examinations).
13. Be willing to signed a written informed consent document before enrollment.

Exclusion Criteria:

1. Patients combined with HAV, HEV, HIV or other infectious diseases.
2. Acute infections, gastrointestinal bleeding, etc. occurred within 30 days before screening.
3. Women who are pregnant (urine/blood pregnancy test positive) or lactating; patients with severe autoimmune diseases; patients with uncontrolled infectious diseases.
4. Major organs dysfunction.
5. Combined with other severe organic diseases or mental illnesses, including any uncontrolled clinically significant systematic diseases such as urinary, circulatory, respiratory, neurological, psychiatric, digestive, endocrine and immune diseases.
6. Allergic constitution, history of allergies to blood products, known to be allergic to test substances.
7. Immunosuppressive or systemic cytotoxic drugs may require within 6 months prior to screening or during the study; 6 months prior to screening accepted other cell therapies including NK, CIK, DC, CTL and stem cell therapy etc.
8. Patients currently participating in other clinical trials who may violate this treatment plan and observations.
9. Those who are unable or unwilling to provide informed consent or who are unable to comply with the research requirements.
10. Any situation that investigators believe the risk of the subjects is increased or results of the trial are disturbed: patients with any serious acute or chronic physical or mental illness, or laboratory abnormalities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-04-26 (Estimated); Primary Completion 2026-04-26 (Estimated); Study Completion 2026-09-26 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation: Incidence of Adverse events (AEs) | up to 60 weeks
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).
Safety evaluation: Dose limited toxicity (DLTs) | up to 60 weeks
  The incidence, characteristic and severity of DLTs will be recorded and assessed.
Safety evaluation: Maximum-tolerated dose (MTD) | up to 60 weeks
  MTD or clinical recommended dose will be recorded and evaluated.
Efficacy evaluation: Objective Response Rate(ORR) | up to 15months
  Objective clinical response will be assessed by investigators
Efficacy evaluation: Duration of Response(DOR) | up to 15months
  The duration of objective response in patients will be recorded until 15months after the start of 1st cycle of treatment
Efficacy evaluation: Progress Free Survival(PFS) | up to 15months
  Observation for progression-free survival (PFS) will be recorded until 15 months after the start of 1st cycle of treatment
Efficacy evaluation: Overall Survival (OS) | up to 15months
  Observation for overall survival l (OS) will be recorded until 15 months after the start of 1st cycle of treatment.

IPD SHARING:
Plan to Share IPD: No